CLINICAL TRIAL: NCT00357916
Title: A Randomized, Controlled Study to Evaluate the Sensitizing Potential of PEP005 Topical Gel (0.01% Concentration) in Healthy Volunteers Using a Repeat Insult Patch Test Design
Brief Title: Study to Determine the Sensitizing Potential of PEP005 Topical Gel in Healthy Volunteers Using a Repeat Insult Patch Test Design
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peplin (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PEP005-005
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: PEP005; Safety

INTERVENTIONS:
Drug: PEP005 Topical Gel (0.01% concentration)

SUMMARY:
To determine the sensitisation potential of PEP005 Topical Gel (0.01% concentration) on normal skin

To evaluate skin irritation

DETAILED DESCRIPTION:
This is a repeat insult patch test study. On treatment days, the investigational product PEP005 Topical Gel (0.01% concentration) and vehicle control will be applied under open conditions to sites on the infrascapular region of the back 3 times weekly for 3 weeks (9 applications in total) during the induction phase. Following a rest period of approximatley 10-14 days, a single challenge application will be performed. Local tolerability will be assessed visually using an ordinal scoring system. If a cutaneous response observed in the challenge phase indicates possible sensitisation, or at the discretion of the investigator, a rechallenge will occur

ELIGIBILITY:
Inclusion Criteria:

1. are healthy males or females (to be confirmed by medical history);
2. are between 18 and 65 years of age;
3. have Fitzpatick skin type I, II, III, or IV
4. are willing to wait 6 hours after product application to shower;
5. in the case of females of childbearing potential, are using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm, or abstinence), have a negative urine pregnancy test at Screening, and submit to a pregnancy test prior to the challenge application;
6. are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events;
7. have acceptable vital signs (ie oral body temperature, blood pressure (systolic and diastolic), and pulse rate) taken and are willing to have them taken at the end of study (EOS, within 7 days of the initial challenge evaluation);
8. complete a medical screening procedure; and
9. read, understand and provide signed informed consent.

Exclusion Criteria:

1. have any visible skin disease at the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction;
2. have Fitzpatrick skin type V or VI;
3. have excessive hair on their back;
4. current drug or alcohol abuse;
5. have a clinically significant illness that may influence the outcome of the study within the 4 weeks prior to and during the study;
6. are not willing to refrain from using topical/systemic analgesics such as aspirin, Aleve, Motrin, Advil, or Nuprin within 72 hours prior to and during the study (occasional use of Tylenol will be permitted);
7. based on the investigator's initial examination should not participate in the study (ie, non compliance, inability to understand the study and give adequate informed consent)
8. are using systemic/locally-acting medications which might counter or influence the study aim during the study and within 2 weeks prior to the beginning of the study (eg, antihistamines, or topical glucocorticosteroids);
9. are using systemic/locally-acting anti-inflammitories which might counter or influence the study aim during the study and within 72 hours prior to the beginning of the study;
10. are females who are pregnant, plan to become pregnant during the study, or are nursing a child;
11. have a known sensitivity or allergy to constituents present in the material being evaluated; and/or
12. have participated in any clinical testing of an investigational drug within 28-days or any clinical patch study within 14-days prior to or are currently participating in any clinical testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To determine the sensitization potential of PEP005 Topical Gel (0.01% concentration) on normal skin.

SECONDARY OUTCOMES:
To evaluate skin irritation

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Dosik, MD, Principal Investigator — TKL Research, Inc.; Peter Welburn, PhD, Study Director — Peplin Operations (Sponsor)
Locations (1):
- TKL Research Inc, Paramus, New Jersey, United States

REFERENCES:
- [Derived] Dosik JS, Damstra M, Udell C, Welburn P. Evaluation of the skin sensitization, photoirritation, and photoallergic potential of ingenol mebutate gel in healthy volunteers. J Clin Aesthet Dermatol. 2014 Apr;7(4):35-42. PMID 24765228